CLINICAL TRIAL: NCT07276373
Title: A Phase 1b/2, Open-Label, Dose-Finding and Proof of Concept Study of Nenocorilant in Combination With Anti-Programmed Cell Death/(Ligand) 1 in Patients With Advanced Solid Malignancies
Brief Title: Two Part Study of Nenocorilant Combined With Nivolumab in Patients With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CORT125236-750
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
Keywords: Advanced Solid Tumors; Solid Tumors; Solid Malignancies
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1a: Nenocorilant 200 mg and Nivolumab (Experimental): Cohort 1a: Patients will receive nenocorilant 200 mg orally under fed conditions once daily, and nivolumab 240 mg IV every 2 weeks. After 3 months of treatment, patients may choose to switch the nivolumab regimen to 480 mg IV every 4 weeks if the nenocorilant nivolumab combination is tolerated.
  Interventions: Drug: Nenocorilant 200 mg; Drug: Nivolumab
- Cohort 1b: Nenocorilant 300 mg and Nivolumab (Experimental): Cohort 1b: Patients will receive nenocorilant 300 mg orally under fed conditions once daily, and nivolumab 240 mg IV every 2 weeks. After 3 months of treatment, patients may choose to switch the nivolumab regimen to 480 mg IV every 4 weeks if the nenocorilant nivolumab combination is tolerated.
  Interventions: Drug: Nenocorilant 300 mg; Drug: Nivolumab
- Cohort 1c: Nenocorilant 400 mg and Nivolumab (Experimental): Cohort 1c: Patients will receive nenocorilant 400 mg orally under fed conditions once daily, and nivolumab 240 mg IV every 2 weeks. After 3 months of treatment, patients may choose to switch the nivolumab regimen to 480 mg IV every 4 weeks if the nenocorilant nivolumab combination is tolerated.
  Interventions: Drug: Nenocorilant 400 mg; Drug: Nivolumab

INTERVENTIONS:
Drug: Nenocorilant 200 mg — Nenocorilant 200 mg will be supplied as 50 and/or 100 mg tablets.
  Other Names: CORT125236
  Arms: Cohort 1a: Nenocorilant 200 mg and Nivolumab
Drug: Nenocorilant 300 mg — Nenocorilant 300 mg will be supplied as 50 and/or 100 mg tablets.
  Other Names: CORT125236
  Arms: Cohort 1b: Nenocorilant 300 mg and Nivolumab
Drug: Nenocorilant 400 mg — Nenocorilant 400 mg will be supplied as 50 and/or 100 mg tablets.
  Other Names: CORT125236
  Arms: Cohort 1c: Nenocorilant 400 mg and Nivolumab
Drug: Nivolumab — Nivolumab 240 mg and 480 mg will be supplied as single-dose 120 mg/12 mL (10 mg/mL) vials.

SUMMARY:
This open-label, dose-finding, and proof of concept study will evaluate the safety, tolerability, maximum-tolerated dose (MTD) and/or optimal dose of nenocorilant when administered in combination with nivolumab in patients with advanced solid malignancies.

DETAILED DESCRIPTION:
This is a Phase 1b/2 study that consists of 2 parts.

In the dose-finding Phase 1b part, researchers will evaluate escalating dose levels of nenocorilant (given with a fixed dose and schedule of nivolumab) in patients with advanced solid malignancies. All patients will be treated with the combination of nenocorilant plus nivolumab in 28-day cycles. Nenocorilant will be administered orally once daily using a continuous dosing schedule, under fed conditions. Nivolumab will be initially given at 240 mg administered intravenously (IV) once every 2 weeks. After 3 months of treatment, patients may choose to switch to a fixed dosing regimen of 480 mg IV once every 4 weeks if they tolerate the combination regimen of nenocorilant plus nivolumab.

The proof-of-concept Phase 2 part of this study is optional and may be added to further evaluate combination treatment in patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

Part 1

* Signed and dated institutional review board (IRB)/ independent ethics committee (IEC)-approved informed consent form (ICF)
* Has solid malignancies that have received all available standard therapies for the specific tumor type or for which no standard therapy exists, unless patient is intolerant of treatment
* Has a life expectancy of ≥ 3 months
* Has evaluable disease based on RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has adequate organ function
* Negative serum or urine pregnancy test for female patients of childbearing potential
* Agreement to use appropriate precautions to avoid pregnancy, unless the patient and/or their sole sexual partner is permanently sterilized

Exclusion Criteria:

Part 1

* Past or current immune-related adverse events (irAEs) due to anti-programmed cell death protein 1 ligand 1 (PD[L]1) therapy that meet any of the following criteria:

  1. Grade ≥ 3
  2. Resulted in discontinuation of anti-PD(L)1 therapy
* Medical history of an autoimmune or inflammatory disease requiring immunosuppressive therapy
* Medical history of adrenal insufficiency
* Has had any major surgery within 4 weeks prior to the first dose of study treatment
* Concurrent treatment with mifepristone or another glucocorticoid receptor (GR) modulator
* Unable to swallow, retain, or absorb oral medication
* Concurrent participation in another interventional clinical trial
* Has toxicities due to prior therapies that are reversible and have not resolved
* Requirement for treatment with prohibited medications, including but not limited to systemic corticosteroids and cytochrome P450(CYP)3A inducers or inhibitors
* Has a known history of severe hypersensitivity to any of the study drugs, or other human/humanized monoclonal antibodies
* Pregnant or lactating patients or female patients expecting to conceive children within the projected duration of the trial
* Has clinically significant uncontrolled condition(s) which, in the opinion of the Investigator, may confound the results of the trial or interfere with the patient's safety or participation
* Known psychiatric disorder that would interfere with trial compliance
* Has infection with HIV, hepatitis C virus, or hepatitis B virus
* Has untreated parenchymal brain metastasis or has uncontrolled central nervous system metastases
* Has a history of another malignancy within 2 years prior to study treatment, unless cured
* Has received prior autologous or allogeneic organ or tissue transplantation
* A QTcF interval >450 msec, a family history of long QT syndrome or unexplained sudden death at young age, or a requirement for use of medication that may prolong the QTc interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients With 1 or More Adverse Event | From first dose of study treatment up to 28 days after final dose, assessed up to 9 months
Number of Patients With 1 or More Serious Adverse Events | From first dose of study treatment up to 28 days after final dose, assessed up to 9 months
Number of Patients With 1 or More Adverse Events Leading to Study Drug Discontinuation | From first dose of study treatment up to final dose, assessed up to 9 months
Percent of Patients who Experience Dose Limiting Toxicity (DLT) | Up to 28 days after initiation of Cycle 1 (each cycle consists of 28 days)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From date of first dose to progressive disease (PD)/confirmed PD using immune Response Evaluation Criteria in Solid Tumors (iRECIST) (iCPD) or death or start of non-protocol-specified new anticancer therapy, assessed up to 8 months
  To evaluate the proportion of patients with measurable disease at baseline who attain a confirmed complete response (CR) or partial response (PR).
Duration of Response (DoR) | Time of first objective response until PD/iCPD or death or start of non-protocol-specified new anticancer therapy, assessed up to 8 months
  To evaluate DoR as the time from the first CR or PR to first documented PD/iCPD or death or start of non-protocol-specified new anticancer therapy, whichever occurs first.
Best Overall Response (BOR) | From first dose until PD/iCPD or death or start of non-protocol-specified anticancer therapy, assessed up to 8 months
  To evaluate BOR as the proportion of patients with a BOR of CR, PR, stable disease (SD), PD, or nonevaluable.
Duration of SD | Date of start of combined treatment until the criteria for PD/iCPD are met, assessed up to 8 months
  To evaluate duration of SD as defined as the time from the start of combination treatment until the criteria for PD/iCPD are met.
Progression-Free Survival (PFS) | Date of first dose until PD/iCPD or death or start of non-protocol-specified new anticancer therapy, assessed up to 8 months
  To evaluate progression-free survival as the time from the first dose of nenocorilant until PD/iCPD or death or start of non-protocol-specified new anticancer therapy, whichever occurs first.
Change from Baseline of Fridericia-Corrected QT (QTcF) Interval | Baseline to End of Treatment, assessed up to 8 months
Area Under the Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24) of Nenocorilant | Cycle 1 Day 15 predose and 1, 2, 3, 4, and 6 hours postdose and Cycle 2 Day 1 predose (each cycle consists of 28 days)
Maximum Observed Plasma Concentration (Cmax) of Nenocorilant | Cycle 1 Day 15 predose and 1, 2, 3, 4, and 6 hours postdose and Cycle 2 Day 1 predose (each cycle consists of 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Jubb, MD, Study Director — Corcept Therapeutics
Locations (2):
- United States (2):
  - Site 01, San Antonio, Texas
  - Site 02, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No